CLINICAL TRIAL: NCT02156960
Title: Changes of Bone Metabolic Markers and Bone Mineral Density After Denosumab and/or Teriparatide Treatment in Japanese Osteoporotic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant Professor, Shinshu University
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Deno-PTH2365
Record Dates: First submitted 2014-05-31; First posted 2014-06-05 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

ARMS (1):
- Denosumab and/or teriparatide treatment (Experimental): Denosumab and/or teriparatide treatment in osteoporotic patients
  Interventions: Drug: Denosumab treatment in osteoporotic patients; Drug: Teriparatide treatment in osteoporotic patients; Drug: Denosumab and teriparatide treatment in osteoporotic patients

INTERVENTIONS:
Drug: Denosumab treatment in osteoporotic patients — To examine the effectiveness of denosumab in osteoporotic patients
Drug: Teriparatide treatment in osteoporotic patients — To examine the effectiveness of teriparatide in osteoporotic patients
Drug: Denosumab and teriparatide treatment in osteoporotic patients — To examine the effectiveness of denosumab and teriparatide in osteoporotic patients

SUMMARY:
It has not been well known about the changes of bone metabolic markers, bone mineral density and other bone-related markers after teriparatide and/or denosumab treatment in Japanese osteoporotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients

Exclusion Criteria:

* none

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Changes of bone mineral density | every 4-6 months
  Bone mineral density will be examined every 4-6 months to evaluate the suitability of the drug.

SECONDARY OUTCOMES:
Changes of bone turnover markers | every 3-6 months
  Bone turnover markers will be examined every 3-6 months to evaluate the suitability of the drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

REFERENCES:
- [Derived] Nakamura Y, Kamimura M, Ikegami S, Mukaiyama K, Uchiyama S, Taguchi A, Kato H. Changes in serum vitamin D and PTH values using denosumab with or without bisphosphonate pre-treatment in osteoporotic patients: a short-term study. BMC Endocr Disord. 2015 Dec 15;15:81. doi: 10.1186/s12902-015-0077-3. PMID 26666998